CLINICAL TRIAL: NCT02720536
Title: Open-label, Multicenter, Single Arm, Phase III Study to Collect Additional Safety and Efficacy Data With Deferasirox Film-coated Tablets in Patients Completing Study CICL670F2201
Brief Title: Extended Evaluation of Deferasirox Film-coated Tablet (FCT) Formulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AIC04
Record Dates: First submitted 2016-03-21; First posted 2016-03-28 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Chronic Iron Overload
Keywords: adult; pediatric,; anemia.; Myelodysplastic Syndrome; Thalassemia; Film coated tablet; ICL670; MDS; Chelation; Deferasirox; Iron overload
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes; Thalassemia; Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deferasirox (Experimental): Treatment will be administered daily for up to 24 months. For each patient the daily dose is calculated based on the patient's actual body weight.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Deferasirox FCT will be provided as 90 mg, 180 mg and 360 mg film-coated tablets for oral use.

SUMMARY:
Extend evaluation of deferasirox film-coated tablet (FCT) formulation

DETAILED DESCRIPTION:
Collection of additional safety and efficacy data with deferasirox film-coated tablet (FCT) in patients who had completed study CICL670F2201

* Provide patients who completed 24 weeks of treatment in the core study, CICL670F2201, the possibility to have additional treatment with the deferasirox FCT.
* Collect additional longer term data on the safety and the tolerability of the deferasirox FCT.
* Collect efficacy data on the deferasirox FCT in reduction or maintenance of iron burden as measured by serum ferritin level.

ELIGIBILITY:
Key Inclusion Criteria for subjects:

* Completed 24-weeks of study treatment as described in the core protocol (CICL670F2201).
* Were deemed to have tolerated deferasirox treatment by the investigator.
* Provided written informed consent/assent before any study-specific procedures were performed. For pediatric patients, consent was obtained from parent(s) or legal patient's representative. Investigators were to have also obtained assent of patients according to local, regional or national guidelines.

Key Exclusion for subjects:

The exclusion criteria followed those described for the core protocol CICl670F2201, which were as follows:

* Creatinine clearance below the contraindication limit in the locally approved prescribing information.
* Serum creatinine > 1.5 × upper limit of normal range (ULN) at Screening
* Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) > 5 × ULN,
* Significant proteinuria
* Patients with significant impaired gastrointestinal function or gastrointestinal disease
* Clinical or laboratory evidence of active Hepatitis B or Hepatitis C
* Patients with psychiatric or addictive disorders
* Patients with a known history of HIV seropositivity (Elisa or Western blot).
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there was an evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* Patients with a history of hypersensitivity to any of the study drug or excipients.
* Patients with significant medical condition that could interfere with the ability to participate in this study
* Patients who were participating in another clinical trial or receiving an investigational drug.
* Patients using prohibited medication,
* Patients with liver disease with severity of Child-Pugh Class B or C.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using effective methods of contraception during dosing of study treatment

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Novartis Investigative Site, Vienna, Austria
- Greece (3):
  - Novartis Investigative Site, Goudi-Athens, GR
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Italy (9):
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Cagliari, ITA
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tartaglione I, Origa R, Kattamis A, Pfeilstocker M, Gunes S, Crowe S, Fagan N, Vincenzi B, Ruffo GB. Two-year long safety and efficacy of deferasirox film-coated tablets in patients with thalassemia or lower/intermediate risk MDS: phase 3 results from a subset of patients previously treated with deferasirox in the ECLIPSE study. Exp Hematol Oncol. 2020 Aug 10;9:20. doi: 10.1186/s40164-020-00174-2. eCollection 2020. PMID 32793403

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients completed study CICL670F2201 (NCT02125877) prior to entry into this study
Period: Overall Study
Arm/Group | Deferasirox
Started | 53
Completed | 34
Not Completed | 19
Not completed — Primary reason (PR) - subject withdrawal | 11
Not completed — PR - pregnancy | 2
Not completed — PR - unsatisfactory therapeutic effect | 2
Not completed — PR - death | 1
Not completed — PR - adverse event | 1
Not completed — PR - abnormal lab value(s) | 1
Not completed — PR- unwilling to comply with procedures | 1

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox
Number analyzed (Participants) | 53
Age, Customized [Number; unit: Participants]
  <18 | 3
  ≥18 - <50 | 46
  ≥ 50 - <65 | 1
  ≥ 65 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 50
  Asian | 1
  Other | 2
Main underlying disease [Number; unit: participants] — Participants with myelodysplastic syndrome (MDS) and transfusion-dependent thalassemia. The very low, low or intermediate risk MDS was to be determined by the Revised International Prognostic Scoring System (IPSS-R) and IPSS-R was to be confirmed by a bone marrow examination within 6 months prior to study entry. MDS with INT risk =MDS with intermediate risk
  participants
    MDS with very low risk as per the IPSS - R | 2
    MDS with low risk as per the IPSS - R | 1
    MDS with INT risk as per the IPSS - R | 1
    Transfusion-dependent thalassemia | 49

OUTCOME MEASURES:

1. Primary Outcome: Overview of Number of Participants With Adverse Events
Description: Numbers represent counts of participants within the categories. An adverse event (AE) was defined as treatment emergent if its onset date is on or after (≥) the first administration of study treatment within this study or events present prior to start of study treatment but increased in severity on or after (≥) the first administration of study treatment within this study but not later than 30 days after the last study treatment in this study
Time Frame: Baseline up to approximately 25 months
Population: Safety analysis set
Measure: Number; unit: number of participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 53
number of participants
  Adverse events (AEs) | 52
  Treatment related AEs | 20
  Severe adverse events | 14
  Treatment related severe adverse events | 2
  Serious adverse events (SAEs) | 13
  Treatment related SAEs | 0
  Fatal SAEs | 1
  Treatment related fatal SAEs | 0
  AEs leading to discontinuation | 4
  Treatment related AEs leading to discontinuation | 2
  AEs leading to dose adjust/interruption | 33
  AEs requiring additional therapy | 4

2. Primary Outcome: Change From Baseline Red Blood Cells (RBC) (10^12 Cells/L) at Month 6 and Month 12
Description: The change from baseline at each time point is calculated only for subjects with a value at baseline and the particular time point. Post = Post baseline, Change = Post - Baseline
Time Frame: Baseline, 6 and 12 months
Population: Safety analysis set - at each timepoint the subjects from the safety analysis set who have a value of the lab parameter of interest at both baseline and the timepoint of interest
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Groups:
- Baseline: Baseline of laboratory value
- Month 6: Change from baseline at month 6
- Month 12: Change from baseline at month 12
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 53 | 42 | 40
10^12 cells/L
  Baseline | 3.753 (0.4909) | 3.733 (0.5016) | 3.746 (0.5071)
  Post | NA (NA) — No post value at baseline | 3.610 (0.5153) | 3.607 (0.5423)
  Change | NA (NA) — No post value at baseline | -0.124 (0.3892) | -0.139 (0.4330)

3. Primary Outcome: Change From Baseline White Blood Cells (WBC) (10^9 Cells/L) at Month 6 and Month 12
Description: as for outcome 2
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 53 | 42 | 40
10^9 cells/L
  Baseline | 9.336 (5.1383) | 9.559 (5.6650) | 9.100 (5.4667)
  Post | NA (NA) — No post value at baseline | 9.090 (4.3712) | 9.007 (4.4385)
  Change | NA (NA) — No post value at baseline | -0.469 (4.0727) | -0.093 (4.5792)

4. Primary Outcome: Change From Baseline Platelets (10^9 Cells/L) at Month 6 and Month 12
Description: as for outcome 2
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 53 | 42 | 40
10^9 cells/L
  Baseline | 330.1 (188.81) | 336.5 (195.97) | 339.4 (196.41)
  Post | NA (NA) — No post value at baseline | 344.2 (190.43) | 361.9 (165.91)
  Change | NA (NA) — No post value at baseline | 7.7 (112.98) | 22.4 (100.72)

5. Primary Outcome: Change From Baseline Serum Creatinine (Umol/L) at Month 6 and Month 12
Description: as for outcome 2
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 53 | 43 | 40
umol/L
  Baseline | 55.1 (16.16) | 54.4 (16.34) | 57.4 (16.91)
  Post | NA (NA) — No post value at baseline | 62.0 (16.17) | 63.5 (16.78)
  Change | NA (NA) — No post value at baseline | 7.6 (9.51) | 6.1 (11.09)

6. Primary Outcome: Change From Baseline Creatinine Clearance (mL/Min) at Month 6 and Month 12
Description: as for outcome 2
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 52 | 41 | 40
mL/min
  Baseline | 131.9 (51.32) | 131.8 (56.98) | 129.6 (50.30)
  Post | NA (NA) — No post value at baseline | 116.0 (48.71) | 119.8 (49.34)
  Change | NA (NA) — No post value at baseline | -15.8 (35.12) | -9.8 (32.74)

7. Primary Outcome: Change From Baseline Alanine Aminotransferase/Serum Glutamic Pyruvic Transaminase (ALT/SGPT) (U/L) at Month 6 and Month 12
Description: as for outcome 2
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 53 | 44 | 40
U/L
  Baseline | 37.4 (31.47) | 39.4 (33.51) | 39.5 (33.32)
  Post | NA (NA) — No post value at baseline | 28.9 (21.12) | 25.9 (19.08)
  Change | NA (NA) — No post value at baseline | -10.5 (29.16) | -13.6 (27.44)

8. Primary Outcome: Change From Baseline Aspartate Aminotransferase/Serum Glutamic Oxaloacetic Transaminase (AST/SGOT) (U/L) at Month 6 and Month 12
Description: as for outcome 2
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 53 | 43 | 39
U/L
  Baseline | 30.7 (24.40) | 32.9 (26.48) | 33.7 (26.67)
  Post | NA (NA) — No post value at baseline | 27.6 (18.81) | 25.2 (12.78)
  Change | NA (NA) — No post value at baseline | -5.3 (21.03) | -8.5 (19.18)

9. Secondary Outcome: Change From Baseline of Serum Ferritin Level (ug/L) at Month 6 and 12
Description: The change from baseline at each time point is calculated only for subjects with a value at baseline and the particular time point. Post = Post baseline, Change = Post - Baseline. A negative change from baseline is regarded as an improvement in this study
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/l
Groups:
- Baseline: Serum ferritin value at baseline
- Month 6: Serum ferritin value at baseline and at month 6
- Month 12: Serum ferritin value at baseline and at month 12
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 53 | 44 | 36
ug/l
  Baseline | 2523.51 (1746.087) | 2614.12 (1781.287) | 2542.76 (1904.087)
  Post | NA (NA) — No values available | 2228.94 (1910.182) | 1924.49 (1839.818)
  Change | NA (NA) — No values available | -385.18 (1038.789) | -618.26 (1054.150)

10. Secondary Outcome: Percentage Relative Change From Baseline of Serum Ferritin (%) at Month 6 and 12
Description: The percentage relative change from baseline at each time point is calculated only for subjects with a value at baseline and the particular time point. Post = Post baseline, Percentage relative change = 100 × ([Post - Baseline] / Baseline). Percentage relative change is calculated for each patient individually and then overall descriptive summary statistics is obtained for subjects with a value at baseline and the particular time point. A negative percentage relative change from baseline is regarded as an improvement in this study
Time Frame: Baseline, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of relative change
Arm/Group | Baseline | Month 6 | Month 12
Number analyzed (Participants) | 53 | 44 | 36
percentage of relative change | NA (NA) — No values available | -18.61 (32.969) | -29.08 (33.056)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 25 months
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Arm/Group | Deferasirox
All-Cause Mortality (participants affected / at risk) | 1/53
Serious Adverse Events (participants affected / at risk) | 13/53
Other Adverse Events (participants affected / at risk) | 48/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=53)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Goitre (Endocrine disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Diverticulitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lymph gland infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Device failure (Product Issues) | 1
Panic attack (Psychiatric disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=53)
Palpitations (Cardiac disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 10
Abdominal pain upper (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 10
Influenza like illness (General disorders) | 5
Pyrexia (General disorders) | 13
Hypertransaminasaemia (Hepatobiliary disorders) | 4
Ear infection (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 7
Influenza (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 7
Respiratory tract infection (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 6
Blood creatinine increased (Investigations) | 4
Urine protein/creatinine ratio increased (Investigations) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 14
Dysuria (Renal and urinary disorders) | 3
Glycosuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 4
Renal colic (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT02720536/SAP_000.pdf
  • Study Protocol (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT02720536/Prot_001.pdf